CLINICAL TRIAL: NCT05225363
Title: A Phase 1 Study to Evaluate TAG72-Targeting Chimeric Antigen Receptor (CAR) T Cells in Patients With Advanced Epithelial Ovarian Cancer
Brief Title: Modified Immune Cells (TAG72-CAR T Cells) for the Treatment of Patients With Platinum Resistant Epithelial Ovarian Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20034; NCI-2021-10838 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20034 (Other: City of Hope Medical Center); P30CA033572 (NIH); R01CA266874 (NIH)
Record Dates: First submitted 2021-12-08; First posted 2022-02-04 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Platinum-Resistant Ovarian Carcinoma
MeSH Terms: interventions — Immunotherapy, Adoptive; Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (TAG72-CAR T cells) (Experimental): Patients receive fludarabine IV and cyclophosphamide IV on days -5 to -3. Patients receive TAG72-CAR T cells IP on day 0.
  Interventions: Biological: Chimeric Antigen Receptor T-cells; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: Chimeric Antigen Receptor T-cells — Receive TAG72-CAR T cells IP
  Other Names: CAR T Cell; CAR T Cells; CAR T-cells; CAR-modified T-cells; CAR-T Cell; CAR-T Cells; Chimeric-antigen Receptor T-lymphocytes
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine — Given IV
  Other Names: Fluradosa

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of TAG72-chimeric antigen receptor (CAR) T cells in treating patients with epithelial ovarian cancer that remains despite treatment with platinum therapy (platinum resistant). T cells are infection fighting blood cells that can kill tumor cells. The T cells given in this study will come from the patient and will have a new gene put in them that makes them able to recognize TAG72, a protein on the surface of tumor cells. These TAG72-specific T cells may help the body's immune system identify and kill TAG72+ cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of TAG72-CAR T cells in participants with recurrent epithelial ovarian cancer (EOC).

II To determine the maximum tolerated dose (MTD). III. To identify the recommended phase 2 dose (RP2D).

SECONDARY OBJECTIVES:

I. Persistence of CAR T cells in blood and peritoneal cavity pre- and 28 days post-infusion.

II. Response based on Immune-Related Response Criteria (irRC). III. Estimate the 6 month progression free survival rate. IV. Estimate median overall survival. V. TAG72 expression on tumor cells by immunohistochemistry (IHC) and/or flow cytometry; VI. Describe the serum cytokine profile pre- and post-CAR T cell infusion to assess potential cytokine release syndrome (CRS) toxicity and CAR T cell effector function.

EXPLORATORY OBJECTIVES:

I. Phenotypes and frequencies of immune cell subsets in the peripheral blood pre- and post- therapy: analysis will include CD4:CD8 ratios, differentiation status (CD62L, CD27, CD45 RA/RO), and exhaustion markers (PD1, Tim3, LAG3), trafficking (CCR7, alpha4beta7), proliferation markers (ki67) and effector functions (cytotoxicity, Th1/Th2 cytokines, and CD107a degranulation) on endogenous and CAR+ T cells.

II. Phenotype of tumor-infiltrating lymphocytes (TILs). III. Gene expression (by RNA-seq) of circulating tumor cells (CTCs). IV. Circulating cell-free deoxyribonucleic acid (cfDNA) in peripheral blood by whole exome sequencing.

V. CAR immunogenicity based on the presence of anti-TAG72 CAR antibodies or T cell mediated immune responses.

OUTLINE: This is a dose-escalation study of TAG72-CAR T cells.

Patients receive fludarabine intravenously (IV) and cyclophosphamide IV on days -5 to -3. Patients receive TAG72-CAR T cells IP on day 0.

After completion of study treatment, patients are followed up at 1, 7, 14, 21, 28, 60 and 90 days, 6, 9, and 12 months, then for up to 15 years.

ELIGIBILITY:
ELIGIBILITY CRITERIA 1.1 Inclusion Criteria

* Participant must have the ability to understand and the willingness to sign a written informed consent.
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies. If unavailable exceptions may be granted with Study PI approval.
* Age > 18 years.
* ECOG Performance status 0 - 2 or KPS ≥70%.
* Documented platinum resistant EOC (defined as disease that has progressed within six months of completing platinum therapy, or lack of response or disease progression while receiving the most recent platinum-based therapy, respectively). Progression may be determined radiographically (not RECIST) or by new onset of malignant pleural effusion. Participant may have at least 1 measurable lesion or disease measured by PCI at the time of surgery.
* Documented TAG72+ (> 1% cells ≥ +1 intensity) tumor expression by IHC (MAb CC49) as evaluated by COH Pathology Core.
* In addition to platinum agents, participant must have received and failed, or have been intolerant to taxanes, liposomal doxorubicin or other agents known to confer clinical benefit. Participants are not required to fail all of these chemotherapy agents if, in the investigator's opinion, they would benefit from treatment on the current protocol.
* No known contraindications to leukapheresis, steroids or tocilizumab.
* Participant of reproductive potential must agree to use acceptable birth control methods throughout study therapy and for 3 months after final dose of study treatment.
* _ANC ≥ 1,000/mm3
* Total serum bilirubin ≤ 1.5 x ULN Patients with Gilbert syndrome may be included if their total bilirubin is < 3.0 x ULN and direct bilirubin ≤ 1.5 x ULN.
* AST < 3 x ULN if liver metastasis: AST < 5 x ULN)
* ALT < 3 x ULN if liver metastasis: ALT < 5 x ULN)
* Participants not receiving therapeutic anticoagulation: INR or aPTT ≤1.5 x ULN
* Creatinine clearance of ≥ 50 mL/min per the Cockcroft-Gault formula
* Cardiac function (12 lead-ECG) without acute abnormalities requiring investigation or intervention
* Left ventricular ejection fraction >40%
* QuantiFERON-TB Gold or equivalent*

1.2 Exclusion Criteria

* Participant has not yet recovered from toxicities of prior therapy.
* Active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition or other agents used in this study.
* History of (non-infectious or COVID-related) pneumonitis that required steroids or current pneumonitis
* Current signs and/or symptoms of bowel obstruction
* History of inflammatory bowel disease
* History of gastrointestinal perforation or symptomatic diverticular disease
* History of intra-abdominal abscess within the past 3 months.
* Patients with known peritoneal adhesions that preclude the placement of an intraperitoneal catheter in the opinion of the surgeon placing the intraperitoneal catheter.
* Participant with clinically significant arrhythmia or arrhythmias not stable on medical management within two weeks of signing the 'Screening/Leukapheresis/Treatment' consent.
* Participant with known history or prior diagnosis of optic neuritis or other immunologic or inflammatory disease affecting the central nervous system, including seizure disorder.
* Known bleeding disorders (e.g., von Willebrand's disease or hemophilia).
* History of stroke or intracranial hemorrhage within 6 months prior to signing the 'Screening/Leukapheresis/Treatment' consent.
* History of other malignancies, except for malignancy surgically resected (or treated with other modalities) with curative intent with no known active disease present for ≥ 3 years, basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin.
* Uncontrolled active infection.
* Active hepatitis B or hepatitis C infection.
* HIV infection.
* Any other condition that would, in the Investigator's judgment, contraindicate the subject's participation in the clinical study due to safety concerns with clinical study procedures.

  o Massive ascites requiring therapeutic paracentesis will not be cause for ineligibility, per se, but will be evaluated on an individual basis. Investigators who have questions regarding assessing ascites are asked to speak with the Principal Investigator.
* Subject has received or plans to receive the following therapy/treatment prior to leukapheresis or lymphodepleting chemotherapy, unless stopped according to the washout requirements:
* Prospective participants who, in the opinion of the Investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2022-05-05 (Actual); Primary Completion 2026-10-05 (Estimated); Study Completion 2027-06-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) | Up to 28 days
  Rates and associated 90% Clopper and Pearson binomial confidence limits will be estimated.
Incidence of adverse events | Up to 1 year post treatment
  Adverse Events are graded using NCI CTCAE v.5.

SECONDARY OUTCOMES:
Persistence of CAR T cells | Up to 28 days post treatment
  Defined as CAR T cells > 0.1% of total CD3 cells by flow-cytometry.
Expansion of CAR T cells | Up to 1 year post treatment
  Max log10 copies/ug of genomic DNA
Response (iRECIST) | Up to 1 year post treatment
  Assessed based on Immune-Related Response Criteria. Rates and associated 90% Clopper and Pearson binomial confidence limits will be estimated.
Overall survival (OS) | Up to 1 year post treatment
  Defined as death from all causes from first treatment date (either lymphodepletion or CAR T cell infusion, as applicable. Kaplan Meier methods will be used to estimate median OS, and graph the results.
Progression-free survival (PFS) | Up to 6 months post treatment
  Defined as survival without biochemical (CA125) or radiographic evidence of disease progression or relapse from first treatment date (either lymphodepletion or CAR T cell infusion, as applicable). Rates and associated 90% Clopper and Pearson binomial confidence limits will be estimated.
Serum cytokine profile | Up to 1 year post treatment
  Serum cytokine profile before and after CAR T cell infusion: to assess potential cytokine release syndrome (CRS) toxicity and CAR T cell effector function, sequential serum samples will be analyzed for Th1/Th2 cytokines (e.g., IL-12, IFNgamma, TNFalpha, IL-10, IL-4, IL-5) by bead array

OTHER OUTCOMES:
Phenotypes and frequencies of immune cell subsets in the peripheral bloodpre- and post-therapy | Up to 1 year post treatment
  Analysis will include CD4:CD8 ratios, differentiation status (CD62L, CD27, CD45 RA/RO), and exhaustion markers (PD1, Tim3, LAG3),trafficking (CCR7, alpha4beta7), proliferation markers (ki67) and effector functions (cytotoxicity, Th1/Th2 cytokines, and CD107a degranulation) on endogenous and CAR+ T cells. Will provide descriptive statistics for exploratory studies. Data will be presented as % of total cells, or as cell/mL blood or peritoneal fluid.
Phenotype of tumor-infiltrating lymphocytes | Up to 1 year post treatment
  Will provide descriptive statistics for exploratory studies.
Gene expression | Up to 1 year post treatment
  Assessed by ribonucleic acid sequencing (RNA-seq) of circulating tumor cells (CTCs). Will provide descriptive statistics for exploratory studies.
Circulating cell-free deoxyribonucleic acid in peripheral blood | Up to 1 year post treatment
  Assessed by whole exome sequencing.
CAR immunogenicity | Up to 1 year post treatment
  Assessed based on the presence of anti-TAG72 CAR antibodies or T cell mediated immune responses.
Microbial changes (Stool) | Up to 1 year post treatment
  Microbial changes in stool associated with CAR T cell therapy

CONTACTS AND LOCATIONS:
Overall Officials: Lorna Rodriguez, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States